CLINICAL TRIAL: NCT03805581
Title: A Phase II Study to Determine the Safety of Defibrotide in Sickle Cell Disease-Related Acute Chest Syndrome
Brief Title: Defibrotide in Sickle Cell Disease-Related Acute Chest Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC-192
Record Dates: First submitted 2018-12-18; First posted 2019-01-15 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Sickle Cell Disease; Acute Chest Syndrome
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Chest Syndrome | interventions — defibrotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Defibrotide 6.25 mg/kg IV q6h
  Interventions: Drug: Defibrotide

INTERVENTIONS:
Drug: Defibrotide — Defibrotide 6.25 mg/kg IV q6h up to 7 days
  Other Names: Defitelio®

SUMMARY:
This study evaluates the safety of defibrotide in subjects with sickle cell disease (SCD)-associated acute chest syndrome (ACS).

ELIGIBILITY:
Inclusion Criteria:

* SCD-associated ACS with the presence of any two or more of the following signs not explained by other etiologies: Fever, Chest pain, Cough, Dyspnea, Tachypnea for age, Pulmonary infiltrate on CXR and/or Chest CT scan, Decreased O2 saturation with or without oxygen supplement;
* Age 2 to 40 years of age;
* Homozygous Hemoglobin S Disease, Hemoglobin SC Disease or Hemoglobin S 0/+ thalassemia;
* Informed consent/assent;
* Consent of patient/parent within ≤72 hours after inpatient admission for SCD-associated ACS.
* Females of childbearing age will have a negative pregnancy test.

Exclusion Criteria:

* Current Grade III or IV hemorrhage;
* Previous hypersensitivity reaction to defibrotide;
* Current systemic anti-coagulant therapy and/or fibrinolytic therapy;
* Consent of patient/parent greater than 72 hours of inpatient admission for SCD-associated ACS;
* No signed informed consent

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with grade III/IV allergic reaction to defibrotide | 30 days
  All patients will be monitored for allergic reaction probably or definitely related to defibrotide administration.
Number of patients with grade III/IV hemorrhage | 30 days
  All patients will be monitored for hemorrhage probably or definitely related to defibrotide.

SECONDARY OUTCOMES:
Number of patients with improvement in clinical signs of Acute Chest Syndrome | 30 days
  Patients will have pre and post treatment assessments with imaging and blood tests to monitor clinical signs of ACS

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States